CLINICAL TRIAL: NCT02636868
Title: A Multinational, Multicenter, Masked, Randomized, Controlled Study to Assess The Safety and Efficacy of Lucinactant for Inhalation in Preterm Neonates 26 to 32 Weeks Gestational Age With Respiratory Distress Syndrome
Brief Title: The Safety and Efficacy of Lucinactant for Inhalation in Premature Neonates 26 to 32 Weeks Gestational Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Windtree Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03-CL-1202
Record Dates: First submitted 2015-11-19; First posted 2015-12-22 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — lucinactant

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aerosolized lucinactant (low dose) (Experimental): Lucinactant for inhalation with nCPAP; up to 2 repeat doses will be allowed if repeat dosing criteria are met.
  Interventions: Drug: Lucinactant delivered via investigational delivery device; Drug: nCPAP
- Aerosolized lucinactant (high dose) (Experimental): Lucinactant for inhalation with nCPAP; up to 2 repeat doses will be allowed if repeat dosing criteria are met.
  Interventions: Drug: Lucinactant delivered via investigational delivery device; Drug: nCPAP
- nasal CPAP (Active Comparator): nCPAP alone
  Interventions: Drug: nCPAP

INTERVENTIONS:
Drug: Lucinactant delivered via investigational delivery device — Lucinactant for inhalation refers to the active investigational agent lucinactant in combination with the investigational delivery device (drug-device combination product)
  Other Names: AEROSURF
  Arms: Aerosolized lucinactant (high dose); Aerosolized lucinactant (low dose)
Drug: nCPAP — Nasal CPAP

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of lucinactant for inhalation administered as an aerosolized dose in two doses to preterm neonates 26 - 32 weeks gestational age who are receiving nasal continuous positive airway pressure (nCPAP) for Respiratory Distress Syndrome (RDS) compared to neonates receiving nCPAP alone.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the safety and efficacy of lucinactant for inhalation in preterm neonates 26 to 32 completed weeks post-menstrual age (PMA). Efficacy and safety are based on clinical evaluations. The endpoints specified are similar to those in Protocols 03-CL-1201 and 03-CL-1401 to allow for potential comparison and pooling of results.

The objective of this study is to evaluate the safety and efficacy of lucinactant for inhalation in conjunction with nCPAP, compared to nCPAP alone, in preterm neonates with RDS, as assessed by the time to and incidence of respiratory failure and/or death due to RDS over the first 72 hours of life, the incidence of bronchopulmonary dysplasia (BPD) at 36 weeks PMA, and change in physiologic parameters (FiO2 and PCO2) over the first 72 hours of life.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF) from legally authorized representative
2. 26 0/7 to 32 6/7 completed weeks gestation PMA
3. Successful implementation of non-invasive support or ventilation within 90 minutes after birth
4. Spontaneous breathing
5. Chest radiograph consistent with RDS
6. Within the first 20 hours after birth requires an nCPAP of 5 to 7 centimeters water (cmH2O) with a fraction of inspired oxygen (FiO2) of ≥ 0.25 (>0.21 for neonates 26-28 weeks PMA) to 0.40 that is clinically indicated for at least 30 minutes to maintain oxygen by pulse oximetry (SpO2) of 90% to 95%. Transient (<10 minutes) FiO2 excursions outside this range do not reset the 30-minute requirement.

Exclusion Criteria:

1. A heart rate that cannot be stabilized above 100 beats per minute (bpm) within 5 minutes of birth
2. Recurrent episodes of apnea requiring positive pressure ventilation (PPV) administered manually or mechanically through any patient interface
3. A 5 minute Apgar score < 5
4. Major congenital malformation(s) or craniofacial abnormalities that preclude the use of nCPAP, diagnosed antenatally or immediately after birth
5. Clinically significant diseases or conditions other than RDS which could potentially interfere with cardiopulmonary function (e.g. congenital heart disease, hydrops fetalis or congenital infection)
6. A known or suspected chromosomal abnormality or syndrome
7. Premature rupture of membranes (PROM) > 3 weeks
8. Hemodynamic instability requiring vasopressors or steroids for hemodynamic support and/or presumed clinical sepsis
9. A need for intubation and/or mechanical ventilation at any time before enrollment into the study
10. The administration (or plan for administration) of any the following:

    * Another investigational agent or investigational medical device
    * Any other surfactant agent
    * Systemic corticosteroids (other than antenatal steroids already received)
11. Presence of air leak (pneumothorax, pneumomediastinum, pneumopericardium, subcutaneous emphysema, or definite evidence of pulmonary interstitial emphysema (PIE)) on the baseline chest radiograph

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 221 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2019-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Simonson, MD, Study Director — Windtree Therapeutics
Locations (54):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Univ. of Arkansas Medical Center, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital of Orange County, Orange, California
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - Christiana Care Health System, Newark, Delaware
  - University of Miami Holtz Children's Hospital, Miami, Florida
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Albany Medical Center, Albany, New York
  - Morgan Stanley Childrens Hospital of New York Presbyterian (CHONY), New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Brody School of Medicine at ECU, Greenville, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Case Western Reserve University (Rainbow Babies Hosp.), Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Women and Infants Hospital, Providence, Rhode Island
  - Baylor University Medical Center, Dallas, Texas
  - Cook Children's Hospital, Fort Worth, Texas
  - Texas Health Harris Methodist Hospital, Fort Worth, Texas
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Sainte Justine Hospital, Montreal, Quebec
- Chile (7):
  - Hospital Dr Sotero Del Rio, Santiago, Region-MetropolitanadeSantiago
  - Hospital Clínico Regional de Concepción Dr Guillermo Grant Benavente, Concepción
  - Hospital San Jose, Santiago
  - Clinica Alamena de Santiago, Santiago
  - Hospital Santiago Oriente Dr Luis Tisné Brousse, Santiago
  - Hospital Clinico de la Pontificia Universidad Catolica de Chile, Santiago
  - Hospital San Juan de Dios, Santiago
- Colombia (3):
  - Fundacion Hospitalaria San Vicente de Paul, Medellín, Antioquia
  - Hospital General de Medellin, Medellín, Antioquia
  - Fundacion Valle Del Lili, Cali, Valle del Cauca Department
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Csolnoky Ferenc Korhaz, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Okato, Miskolc
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
- Ireland (2):
  - Cork University Hospital, Cork
  - Mid-Western Regional Hospital Limerick, Limerick
- Erasmus Medical Center, Rotterdam, Netherlands
- Poland (9):
  - Ginekologiczno-Polozniczy Szpital Klinicznym UM im. Karola Marcinkowskiego w Poznan i u Katedra Neonatologii, Poznan, Greater Poland Voivodeship
  - S.U. nr2im. Dr. Jana Biziela Oddzial Kliniczny N. W. Z. Intensywna Terapia Noworodka wraz z Wgjazdowy m Zespolem N, Bydgoszcz, Kujawsko-pomorksie
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Oddzial Neonatologii, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Szpital Kliniczny im. Ks, Anny Mazowieckiej Klinika Neonatologii, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Szpital Spegialistycszny nr 2 w Bytomia Oddzial Noworodkow Blok V, Bytom, Silesian Voivodeship
  - Samodzielny Publiczny Specjalistczny Zaklad Opieki Zdrowotnej Zdroje, Szczecin, West Pomeranian Voivodeship
  - Instytut Centrum Zdrowja Matki Polki Klinika Neonatologii, Lodz, Łódź Voivodeship

RESULTS

PARTICIPANT FLOW:
Groups:
- Aerosolized Lucinactant (40 mg TPL/kg); Aerosolized Lucinactant (80 mg TPL/kg): Lucinactant for inhalation with nCPAP; up to 2 repeat doses will be allowed if repeat dosing criteria are met.
  Lucinactant delivered via investigational delivery device: Lucinactant for inhalation refers to the active investigational agent lucinactant in combination with the investigational delivery device (drug-device combination product)
  nCPAP: Nasal CPAP
- nCPAP Only: nCPAP alone
  nCPAP: Nasal CPAP
Period: Overall Study
Arm/Group | Aerosolized Lucinactant (40 mg TPL/kg) | Aerosolized Lucinactant (80 mg TPL/kg) | nCPAP Only
Started | 73 | 76 | 72
Completed | 73 | 75 | 70
Not Completed | 0 | 1 | 2
Not completed — Death | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerosolized Lucinactant (40 mg TPL/kg) | Aerosolized Lucinactant (80 mg TPL/kg) | nCPAP Only | Total
Number analyzed (Participants) | 73 | 76 | 72 | 221
Age, Customized [Mean (Standard Deviation); unit: weeks post menstrual age]
  Gestational Age | 30.8 (1.24) | 30.7 (1.17) | 30.7 (1.17) | 30.7 (1.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 39 | 37 | 107
  Male | 42 | 37 | 35 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 24 | 18 | 61
  Not Hispanic or Latino | 54 | 52 | 54 | 160
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 6 | 16
  White | 62 | 64 | 58 | 184
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 7 | 19
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 2 | 3 | 9
  Colombia | 4 | 7 | 5 | 16
  Netherlands | 2 | 1 | 2 | 5
  Hungary | 6 | 3 | 9 | 18
  United States | 20 | 25 | 21 | 66
  Ireland | 1 | 2 | 0 | 3
  Poland | 23 | 21 | 21 | 65
  Chile | 13 | 15 | 11 | 39
Birth Weight [Mean (Standard Deviation); unit: grams] | 1557.0 (342.38) | 1505.8 (378.5) | 1446.4 (359.13) | 1503.4 (361.73)
Ruptured Membranes [Count of Participants; unit: Participants]
  Spontaneous | 23 | 16 | 19 | 58
  Artificial | 50 | 60 | 53 | 163
Chorioamnionitis [Count of Participants; unit: Participants]
  Yes | 3 | 3 | 2 | 8
  No | 70 | 73 | 70 | 213
Steroid Use, Maternal [Count of Participants; unit: Participants]
  Used Steroids | 68 | 69 | 70 | 207
  No Steroids | 5 | 7 | 2 | 14
Mode of Delivery [Count of Participants; unit: Participants]
  Vaginal | 17 | 12 | 16 | 45
  Cesarean Section | 56 | 64 | 56 | 176
Birth Status [Count of Participants; unit: Participants]
  Single Birth | 44 | 53 | 50 | 147
  Multiple Birth | 29 | 23 | 22 | 74
Appearance, Pulse, Grimace, Activity, and Respiration (Apgar) Score at One Minute [Mean (Standard Deviation); unit: Scores on a scale] — In the test, five things are used to check a baby's health at 1 minutes after birth. Each is scored on a scale of 0 to 2, with 2 being the best score:
  Appearance (skin color) Pulse (heart rate) Grimace response (reflexes) Activity (muscle tone) Respiration (breathing rate and effort) The individual scores are summed to determine the total score.
  Scores on a scale | 6.7 (1.74) | 6.5 (1.71) | 6.8 (1.61) | 6.6 (1.69)
Apgar Score at Five Minutes [Mean (Standard Deviation); unit: Scores on a scale] — In the test, five things are used to check a baby's health at 5 minutes after birth. Each is scored on a scale of 0 to 2, with 2 being the best score:
  Appearance (skin color) Pulse (heart rate) Grimace response (reflexes) Activity (muscle tone) Respiration (breathing rate and effort) The individual scores are summed to determine the total score.
  Scores on a scale | 8.1 (0.90) | 8.0 (1.02) | 8.1 (1.00) | 8.1 (0.97)
Congenital Anomaly [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 0 | 1
  No | 72 | 76 | 72 | 220

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Respiratory Failure or Death Due to Respiratory Distress Syndrome (RDS)
Description: Number of participants who had respiratory failure due to RDS or death due to RDS; known as nasal continuous positive airway pressure (nCPAP) failure
Time Frame: 72 hours
Population: Modified Intent-to-Treat; randomized subjects who received study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Aerosolized Lucinactant (40 mg TPL/kg) | Aerosolized Lucinactant (80 mg TPL/kg) | nCPAP Only
Number analyzed (Participants) | 70 | 72 | 71
Participants | 31 | 32 | 31
Statistical Analysis 1: Comparison: Aerosolized Lucinactant (40 mg TPL/kg) vs Aerosolized Lucinactant (80 mg TPL/kg) vs nCPAP Only; Null hypothesis is no difference across treatment groups; Test type: Superiority; p = 0.363, Regression, Logistic — a priori threshold of statistical significance set at 0.05; Pooled site, treatment, gender, birth weight, and baseline fraction of inspired oxygen (FiO₂) in model
Statistical Analysis 2: Comparison: Aerosolized Lucinactant (40 mg TPL/kg) vs nCPAP Only; Null hypothesis of no difference between treatments; Test type: Superiority; p = 0.360, Regression, Logistic — a priori threshold of statistical significance set at 0.05; Pooled site, treatment, gender, birth weight, and baseline FiO₂ in model
Statistical Analysis 3: Comparison: Aerosolized Lucinactant (80 mg TPL/kg) vs nCPAP Only; Null hypothesis of no difference between treatments; Test type: Superiority; p = 0.461, Regression, Logistic — a priori threshold of statistical significance set at 0.05; Pooled site, treatment, gender, birth weight, and baseline FiO₂ in model

2. Secondary Outcome: Incidence of Respiratory Failure or Death Due to RDS
Description: Incidence of Respiratory Failure or Death Due to RDS by Intubation or Failure Criteria
Time Frame: 72 hours
Population: Modified Intent-to-Treat Population without Treatment Interruptions
Measure: Count of Participants; unit: Participants
Arm/Group | Aerosolized Lucinactant (40 mg TPL/kg) | Aerosolized Lucinactant (80 mg TPL/kg) | nCPAP Only
Number analyzed (Participants) | 64 | 44 | 71
Participants | 28 | 14 | 31
Statistical Analysis 1: Comparison: Aerosolized Lucinactant (40 mg TPL/kg) vs Aerosolized Lucinactant (80 mg TPL/kg) vs nCPAP Only; Null hypothesis is no difference across treatment groups; Test type: Superiority; p = 0.401, Regression, Logistic — a priori threshold of statistical significance set at 0.05; Pooled site, treatment, gender, birth weight, and baseline FiO₂ in model
Statistical Analysis 2: Comparison: Aerosolized Lucinactant (40 mg TPL/kg) vs nCPAP Only; Null hypothesis is no difference across treatment groups; Test type: Superiority; p = 0.372, Regression, Logistic — a priori threshold of statistical significance set at 0.05; Pooled site, treatment, gender, birth weight, and baseline FiO₂ in model
Statistical Analysis 3: Comparison: Aerosolized Lucinactant (80 mg TPL/kg) vs nCPAP Only; Null hypothesis is no difference across treatment groups; Test type: Superiority; p = 0.648, Regression, Logistic — a priori threshold of statistical significance set at 0.05; Pooled site, treatment, gender, birth weight, and baseline FiO₂ in model

3. Secondary Outcome: Time to nCPAP Failure
Description: Time from birth to nCPAP Failure
Time Frame: 72 hours
Population: Modified Intent-to-Treat; randomized participants who received study treatment
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Aerosolized Lucinactant (40 mg TPL/kg) | Aerosolized Lucinactant (80 mg TPL/kg) | nCPAP Only
Number analyzed (Participants) | 70 | 72 | 71
hours | 39.3 (2.06) | 44.8 (2.69) | 40.7 (2.44)
Statistical Analysis 1: Comparison: Aerosolized Lucinactant (40 mg TPL/kg) vs Aerosolized Lucinactant (80 mg TPL/kg) vs nCPAP Only; Null hypothesis of no difference across treatments; Test type: Superiority; p = 0.996, Log Rank — a priori threshold of statistical significance set at 0.05
Statistical Analysis 2: Comparison: Aerosolized Lucinactant (40 mg TPL/kg) vs nCPAP Only; Null hypothesis of no difference between treatments; Test type: Superiority; p = 0.951, Log Rank — a priori threshold of statistical significance set at 0.05
Statistical Analysis 3: Comparison: Aerosolized Lucinactant (80 mg TPL/kg) vs nCPAP Only; Null hypothesis of no difference between treatments; Test type: Superiority; p = 0.995, Log Rank — a priori threshold of statistical significance set at 0.05

4. Secondary Outcome: Incidence of Respiratory Failure or Death Due to RDS With Poisson Distribution Modeling
Description: The measure tests the differences between treatments on respiratory failure or death due to RDS using Poisson distribution modeling, which accounts for the time over which the event could have occurred.
Time Frame: 72 hours
Population: Modified Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Aerosolized Lucinactant (40 mg TPL/kg) | Aerosolized Lucinactant (80 mg TPL/kg) | nCPAP Only
Number analyzed (Participants) | 70 | 72 | 71
Participants | 31 | 32 | 31
Statistical Analysis 1: Comparison: Aerosolized Lucinactant (40 mg TPL/kg) vs Aerosolized Lucinactant (80 mg TPL/kg) vs nCPAP Only; Null hypothesis of no difference between treatment groups; Test type: Superiority; p = 0.312, Regression, Linear — A priori threshold of statistical significance set at 0.10; Generalized linear model using Poisson distribution with pooled site, treatment, gender, birth weight, and baseline FiO₂ in model
Statistical Analysis 2: Comparison: Aerosolized Lucinactant (40 mg TPL/kg) vs nCPAP Only; Null hypothesis of no difference between treatment groups; Test type: Superiority; p = 0.094, Regression, Linear — A priori threshold of statistical significance set at 0.10; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Aerosolized Lucinactant (80 mg TPL/kg) vs nCPAP Only; Null hypothesis of no difference between treatment groups; Test type: Superiority; p = 0.414, Regression, Linear — A priori threshold of statistical significance set at 0.10; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Incidence of Respiratory Failure or Death Due to RDS
Description: Incidence of Respiratory Failure or Death due to RDS by Intubation or Failure Criteria
Time Frame: 28 days
Population: Modified Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Aerosolized Lucinactant (40 mg TPL/kg) | Aerosolized Lucinactant (80 mg TPL/kg) | nCPAP Only
Number analyzed (Participants) | 70 | 72 | 71
Participants | 35 | 32 | 31
Statistical Analysis 1: Comparison: Aerosolized Lucinactant (40 mg TPL/kg) vs Aerosolized Lucinactant (80 mg TPL/kg) vs nCPAP Only; Null hypothesis of no difference between treatment groups; Test type: Superiority; p = 0.099, Regression, Logistic — A priori statistical significance of 0.05; Pooled site, treatment, gender, birth weight, and baseline fraction of inspired oxygen (FiO2) in model
Statistical Analysis 2: Comparison: Aerosolized Lucinactant (40 mg TPL/kg) vs nCPAP Only; Null hypothesis of no difference between treatments; Test type: Superiority; p = 0.090, Regression, Logistic — A priori statistical significance of 0.05; Pooled site, treatment, gender, birth weight, and baseline FiO2 in model
Statistical Analysis 3: Comparison: Aerosolized Lucinactant (80 mg TPL/kg) vs nCPAP Only; Null hypothesis of no difference between treatment groups; Test type: Superiority; p = 0.461, Regression, Logistic — A priori statistical significance of 0.05; Pooled site, treatment, gender, birth weight, and baseline FiO2 in model

6. Secondary Outcome: Number of Participants With Bronchopulmonary Dysplasia (BPD)
Description: Summarizes the number of participants with BPD or alive without BPD
Time Frame: 36 weeks post-menstrual age (PMA)
Population: Modified Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Aerosolized Lucinactant (40 mg TPL/kg) | Aerosolized Lucinactant (80 mg TPL/kg) | nCPAP Only
Number analyzed (Participants) | 70 | 72 | 71
Participants
  BPD | 7 | 7 | 10
  Alive without BPD | 62 | 64 | 59
Statistical Analysis 1: Comparison: Aerosolized Lucinactant (40 mg TPL/kg) vs Aerosolized Lucinactant (80 mg TPL/kg) vs nCPAP Only; Null hypothesis of no treatment between treatments; Test type: Superiority; p = 0.534, ANOVA — A priori threshold for statistical significance set at 0.05; treatment and pooled site in model
Statistical Analysis 2: Comparison: Aerosolized Lucinactant (80 mg TPL/kg) vs nCPAP Only; Null hypothesis of no difference between treatment groups; Test type: Superiority; p = 0.480, ANOVA — A priori threshold for statistical significance set at 0.05; Treatment and pooled site in model
Statistical Analysis 3: Comparison: Aerosolized Lucinactant (80 mg TPL/kg) vs nCPAP Only; Null hypothesis of no difference between treatment groups; Test type: Superiority; p = 0.313, ANOVA — A priori threshold for statistical significance set at 0.05; Treatment and pooled site in model

ADVERSE EVENTS:
Time Frame: Enrollment to 36 weeks post-menstrual age
Arm/Group | Aerosolized Lucinactant (40 mg TPL/kg) | Aerosolized Lucinactant (80 mg TPL/kg) | nCPAP Only
All-Cause Mortality (participants affected / at risk) | 0/70 | 1/72 | 2/71
Serious Adverse Events (participants affected / at risk) | 16/70 | 14/72 | 20/71
Other Adverse Events (participants affected / at risk) | 65/70 | 69/72 | 66/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerosolized Lucinactant (40 mg TPL/kg) (N=70) | Aerosolized Lucinactant (80 mg TPL/kg) (N=72) | nCPAP Only (N=71)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Patent ductus arteriosus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coarctation of the aorta (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neurological infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nocosomial infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis neonatal (Infections and infestations) | 2 (3) | 3 (3) | 5 (6)
Septic embolus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intraventricular haemorrhage neonatal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 1 (1)
Necrotising enterocolitis neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Neonatal respiratory distress syndrome (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 2 (2) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Apnoea neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 7 (8)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary interstitial emphysema syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Pulmonary oedema neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerosolized Lucinactant (40 mg TPL/kg) (N=70) | Aerosolized Lucinactant (80 mg TPL/kg) (N=72) | nCPAP Only (N=71)
Anaemia neonatal (Blood and lymphatic system disorders) | 22 (26) | 31 (37) | 31 (52)
Coagulation disorder neonatal (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 6 (6) | 5 (5)
Patent ductus arteriosus (Cardiac disorders) | 18 (18) | 24 (24) | 24 (26)
Tachycardia (Cardiac disorders) | 6 (6) | 6 (9) | 2 (2)
Atrial septal defect (Congenital, familial and genetic disorders) | 4 (5) | 4 (4) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 6 (7) | 5 (8) | 6 (8)
Constipation (Gastrointestinal disorders) | 6 (7) | 9 (9) | 6 (7)
Gastric haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2) | 6 (6)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 1 (1) | 4 (4) | 4 (4)
Regurgitation (Gastrointestinal disorders) | 10 (10) | 12 (13) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (9) | 9 (10) | 8 (9)
Oedema (General disorders) | 7 (7) | 5 (7) | 7 (7)
Conjunctivitis (Infections and infestations) | 4 (5) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 4 (4) | 1 (1)
Sepsis neonatal (Infections and infestations) | 2 (2) | 3 (3) | 8 (8)
Cardiac murmur (Investigations) | 5 (5) | 4 (4) | 1 (1)
Oxygen saturation decreased (Investigations) | 22 (31) | 25 (35) | 15 (22)
Feeding intolerance (Metabolism and nutrition disorders) | 11 (11) | 17 (17) | 10 (11)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 3 (3)
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 4 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (4) | 7 (7) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1) | 3 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (7) | 6 (6) | 5 (6)
Metabolic acidosis (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 9 (11)
Agitation neonatal (Pregnancy, puerperium and perinatal conditions) | 7 (8) | 9 (10) | 3 (3)
Bradycardia neonatal (Pregnancy, puerperium and perinatal conditions) | 6 (7) | 8 (8) | 3 (3)
Intraventricular haemorrhage neonatal (Pregnancy, puerperium and perinatal conditions) | 7 (8) | 10 (11) | 12 (15)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 41 (47) | 49 (50) | 41 (46)
Neonatal respiratory distress syndrome (Pregnancy, puerperium and perinatal conditions) | 10 (12) | 8 (8) | 13 (13)
Retinopathy of prematurity (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 6 (6) | 3 (3)
Weight decrease neonatal (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 4 (4) | 2 (2)
Apnoea neonatal (Respiratory, thoracic and mediastinal disorders) | 31 (39) | 26 (29) | 27 (31)
Atelectasis neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 4 (5)
Bronchopulmonaria dysplasia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6) | 9 (9)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (10) | 7 (7)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 10 (11) | 8 (9)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (7) | 2 (2)
Hypotension (Vascular disorders) | 2 (3) | 4 (4) | 3 (4)
Pallor (Vascular disorders) | 10 (11) | 4 (5) | 3 (3)

LIMITATIONS AND CAVEATS:
Clogging of a in-line filter led to a higher number of treatment interruptions than expected. This primarily affected one batch of supplies that were, by chance, predominantly used in European sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Steering Committee is responsible for publications, including who will be authoring publications. The sponsor has the right to review publications before they are published and can provide suggested edits, but cannot require changes or prevent publication.

DOCUMENTS (3):
  • Study Protocol (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT02636868/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT02636868/SAP_001.pdf
  • Informed Consent Form (2016-02-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT02636868/ICF_002.pdf